CLINICAL TRIAL: NCT05175261
Title: Assessment of Individual Risk of Cardiovascular Events by Platelet FcGammaRIIa
Status: Completed | Type: Observational
Sponsor: Prolocor, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: PRL-0001
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: STEMI; NSTEMI
Keywords: biomarker; platelet; prognosis; cardiovascular
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Prolocor pFCG test — Perform pFCG test on patients admitted with myocardial infarction to assess prognosis

SUMMARY:
This is a Prospective, Observational Multicenter Non-Interventional Cohort Study. The primary objective is to determine whether platelet expression of FcγRIIa is associated with risk of myocardial infarction (MI), stroke and death. Secondary objectives include: 1) Develop a score that combines clinical characteristics plus platelet expression of FcγRIIa to determine the risk of MI, stroke, and death; and 2) Determine whether platelet expression of FcγRIIa is associated with risk of major bleeding. The primary endpoint is the composite of death, MI and stroke. A secondary endpoint is the incidence of clinically significant bleeding according to the Bleeding Academic Research Consortium (BARC) scale type 2-5. Approximately 800 male and female subjects with confirmed MI [ST-segment elevation MI (STEMI) or non-ST-segment elevation MI (NSTEMI)] will be enrolled before hospital discharge for the index event. Approximately 10 sites in the United States will participate in this study. It is anticipated that it will take approximately 12 months to enroll approximately 800 subjects. The study and subject follow-up will continue until 1) at least 80 ischemic events (MI, stroke, and death) have occurred, and 2) the last subject enrolled has completed 18 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 Myocardial Infarction (STEMI and NSTEMI)
2. Must have ≥ 2 of the following risk factors:

   1. Age ≥ 65
   2. Multi-vessel coronary artery disease (MVD) defined as ≥2 vessels or left main with a stenosis ≥50%
   3. Chronic kidney disease (CKD) defined as estimated glomerular filtration rate (GFR) ˂ 60 mL/min/1.73 m2
   4. Diabetes mellitus (DM)
   5. Prior MI
3. Must agree to participate in the study, to comply with all study procedures and follow-up contact
4. Signed the informed consent form

Exclusion Criteria:

1. Requirement for treatment with full dose anticoagulant therapy (e.g., for atrial fibrillation)
2. Participation in another trial in which the subject is known to receive or could receive anticoagulant or antiplatelet treatment as part of the trial intervention.
3. Non-cardiovascular conditions that, in the judgment of the investigator, will limit survival to less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 800 male and female subjects with confirmed MI [ST-segment elevation MI (STEMI) or non-ST-segment elevation MI (NSTEMI)] will be enrolled before hospital discharge for the index event.
Sampling Method: Non-Probability Sample
Enrollment: 764 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Schneider, MD, Principal Investigator — Prolocor, Inc
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schneider DJ, McMahon SR, Angiolillo DJ, Fanaroff AC, Ibrahim H, Hohl PK, Wanamaker BL, Effron MB, DiBattiste PM; Investigators. Predictive Value of Platelet FcgammaRIIa in Patients Treated With PCI Compared With Medical Therapy Alone After Myocardial Infarction. Circ Cardiovasc Interv. 2025 Apr;18(4):e014939. doi: 10.1161/CIRCINTERVENTIONS.124.014939. Epub 2025 Mar 26. PMID 40135363
- [Result] Schneider DJ, McMahon SR, Angiolillo DJ, Fanaroff A, Ibrahim H, Hohl PK, Wanamaker BL, Effron MB, DiBattiste PM. Platelet FcgammaRIIa as a Marker of Cardiovascular Risk After Myocardial Infarction. J Am Coll Cardiol. 2024 Oct 29;84(18):1721-1729. doi: 10.1016/j.jacc.2024.08.051. PMID 39443015

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Myocardial Infarction: Adults (age>18) were enrolled in this prospective observational non-interventional study after providing written informed consent. Patients were enrolled during hospitalization for type 1 MI (ST elevation or non-ST elevation). Most commonly, patients were enrolled shortly before discharge after therapeutic interventions were completed and clinical judgment was used to determine whether the MI was type 1. Inclusion criteria required that participants had at least 2 of the following: age ≥ 65, multi-vessel coronary artery disease, prior MI, chronic kidney disease (defined as glomerular filtration rate (GFR) ˂60 ml/min/1.73 m2), or diabetes mellitus. These criteria were used to target a higher risk patient group that would have an estimated risk of ~10% for the composite endpoint of MI, stroke, and death (15). This study focused on patients treated with antiplatelet therapy, however, a limited number (n = approximately 100) of patients treated with long term anticoagulants were permitted. Patients were excluded if they were enrolled in another trial in which the subject could receive anticoagulant or antiplatelet treatment as part of the trial intervention; and when non-cardiovascular conditions, in the judgment of the investigator, would limit survival to less than 2 years.
Period: Overall Study
Arm/Group | Patients With Myocardial Infarction
Started | 764
Completed | 757
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Myocardial Infarction
Number analyzed (Participants) | 764
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 197
  >=65 years | 567
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245
  Male | 519
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 17
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 98
  White | 595
  More than one race | 50
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Ischemic
Description: compare the hazard ratio for first occurrence of myocardial infarction (MI), stroke and death in patients with high vs low platelet FcGammaRIIa
Time Frame: Study Duration (up to 3 years)
Measure: Number (95% Confidence Interval); unit: Hazard Ratio comparing high and low pFCG
Arm/Group | Patients With Myocardial Infarction
Number analyzed (Participants) | 567
Hazard Ratio comparing high and low pFCG
  MI, stroke, and death | 2.09 [1.34 to 3.26]
  MI and death | 2.71 [1.73 to 4.25]
  MI | 3.24 [1.64 to 6.37]
  death | 2.57 [1.5 to 4.4]

2. Secondary Outcome: Risk Score
Description: • Develop a score that combines clinical characteristics plus platelet expression of FcγRIIa to determine the risk of MI, stroke, and death
Time Frame: Study Duration (up to 3 years)
Reporting Status: Not Posted

3. Secondary Outcome: Bleeding
Description: compare the hazard ratio for first occurrence of bleeding (bleeding academic research consortium 2, 3, and 5) in patients with high vs low platelet FcGammaRIIa
Time Frame: Study Duration (up to 3 years)
Measure: Number (95% Confidence Interval); unit: Hazard Ratio comparing high and low pFCG
Arm/Group | Patients With Myocardial Infarction
Number analyzed (Participants) | 764
Hazard Ratio comparing high and low pFCG | 1.84 [0.96 to 4.06]

ADVERSE EVENTS:
Time Frame: Adverse events were collected through study completion, an average of 21 months
Description: Myocardial infarction, stroke, bleeding, and death were study endpoints and so were not considered adverse events.
Arm/Group | Patients With Myocardial Infarction
All-Cause Mortality (participants affected / at risk) | 22/764
Serious Adverse Events (participants affected / at risk) | 0/764
Other Adverse Events (participants affected / at risk) | 0/764

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT05175261/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT05175261/SAP_001.pdf